CLINICAL TRIAL: NCT04638257
Title: A Phase I, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Effects of Probiotic Lactobacilli on Vaginal Flora of Pregnant Women
Brief Title: Role of Oral Lactobacilli on Vaginal Flora of Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-239
Record Dates: First submitted 2015-10-05; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacilli (Experimental): Lactobacilli rhamnosus GR-1 and Lactobacilli fermentum RC-14 Lactobacilli rhamnosus GR-1 and Lactobacilli fermentum RC-14
  Interventions: Biological: Lactobacilli rhamnosus GR-1 and Lactobacilli fermentum RC-14
- Placebo (Placebo Comparator): Receives placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Lactobacilli rhamnosus GR-1 and Lactobacilli fermentum RC-14 — Daily oral Lactobacilli starting at =<18 weeks of gestation in singleton pregnancy
  Arms: Lactobacilli
Other: Placebo — Daily oral placebo starting at =<18 weeks of gestation in singleton pregnancy
  Arms: Placebo

SUMMARY:
Bacterial vaginosis (BV) occurs in about 20% of pregnancies and responsible for up to 25% of visits to gynecological clinics. BV is characterized by a shift in vaginal bacterial flora from lactobacilli to pathogenic bacterial flora like Gardnerella and Mycoplasma. Risk factors for the development of BV include douching, use of intrauterine contraceptive devices, new or multiple sexual partners, smoking and African American background.

DETAILED DESCRIPTION:
Diagnosis of BV based on Amsel's criteria and Nugent's scoring. In Amsel's criteria include: presence of thin vaginal discharge, clue cells, vaginal fluid pH >4.5 and positive whiff test. The Nugent score is derived from gram-stained vaginal smear; yielding a score between 0 - 10. A score of, 4 is normal, 4 - 6 is intermediate and a score >7 represents BV. CDC recommends diagnosis of BV on the presence of >3 Amsel criteria and a Nugent score >7. FDA recommends, verification of BV cure should be conducted 21 - 30 days after the initiation of therapy (absence of Amsel's criteria and Nugent score <4).

Cure rate of BV with conventional anti-microbial agents have been disappointing due to high recurrence rate of BV. Recurrence of BV results in repeated exposure to anti-microbial agents which may lead to emergence of drug-resistance strains & the potential for adverse reactions. This suggests a need for alternative therapeutic measures of BV.

Lactobacilli rhamnosus GR-1 and Lactobacilli fermentum RC-14 are H2O2 producing lactobacilli which are toxic to bacteria causing BV by antagonizing the growth and adhesion of pathologic bacteria causing BV. In non-pregnant women, oral administrations of these strains of lactobacilli are safe, and reduce the risk of BV by restoring predominant lactobacilli, the normal vaginal bacterial flora.

Bacterial vaginosis is associated with increased incidence of preterm delivery. For pregnant women, restoration of lactobacilli in the genital tract could be very important to prevent BV and may lower the risk of preterm labor. At present, the safety, tolerability and efficacy of lactobacilli use during pregnancy is not well known for the fetus and the pregnant women. The investigators plan to do a phase I trial to evaluate the safety, tolerability, and efficacy of oral lactobacilli on vaginal flora of pregnant women and follow up their infants for any side effect up to 6 months of age.

In summary, treatment failure and recurrence of BV following anti-microbial treatment is frustrating. During pregnancy, probiotics may be the next step to treat BV and restore normal vaginal micro flora. But the safety of lactobacilli use during pregnancy is not established. The investigators will do phase I trial to evaluate safety of oral lactobacilli in pregnant women along with their infants up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women <18 weeks gestational age
2. >18 years old and able provide informed consent
3. No clinical bacterial vaginosis requiring anti-microbial treatment
4. BV Blue test positive on screening
5. Planned or probable delivery at UTMB, Galveston

Exclusion Criteria:

1. Taking antibiotics or any other microbial at the time of recruitment
2. Documented need for cervical cerclage
3. Multi fetal pregnancy
4. Known aneuploidy or lethal fetal anomalies
5. Illicit drug use
6. Serious maternal medical conditions

   1. Renal insufficiency with serum creatinine >1.5, known proteinuria >300mg/24 hours or receiving dialysis.
   2. Chronic liver disease with liver transaminases >2 times the upper limit of the normal range
   3. Organ transplant recipients.
   4. Severe pulmonary disorder (such as significant obstructive/restrictive disorder, pulmonary hypertension, cystic fibrosis, and chronic oxygen requirement).
   5. Severe heart disease (such as cardiomyopathy with decreased left ventricular ejection fraction, obstructive valvular disease, replaced heart valve, uncorrected aortic coarctation or tetrology).
   6. Established lupus anticoagulant syndrome or antiphospholipid syndrome).
   7. Diabetes class C and greater
   8. Chronic conditions requiring medications for control (such as chronic hypertension, SLE, inflammatory bowel disease, and asthma).
   9. Acquired Immunodeficiency Syndrome or HIV infection without AIDS.
7. Medical complications of pregnancy

   1. Pre-eclampsia
   2. Thrombophilia
   3. Pregnancy induced hypertension
   4. Gestational diabetes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Pregnancy (<18 weeks gestation) for 60 days
  This number will determine if oral supplementation of lactobacilli is safe and tolerated by pregnant women.

SECONDARY OUTCOMES:
Number of participants with incidence and severity of Bacterial Vaginosis during pregnancy assessing for positive lab results screening for Bacterial Vaginiosis | baseline up until 8 (after starting the study drug)
  1. BV Blue test
  2. Nugent scoring
  3. Amsel clinical criteria
Number of Preterm deliveries | baseline up until 36 weeks gestation
  Preterm delivery (<37 weeks gestation)
Measure the inflammatory markers in the vaginal secretions | baseline up until 8 (after starting the study drug)
  1. IL1β
  2. IL6
  3. IL8
  4. TNF-α
  5. GmCSF

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K Jain, MD, Principal Investigator — The University of Texas Medical Branch, Galveston

IPD SHARING:
Plan to Share IPD: No